CLINICAL TRIAL: NCT05226156
Title: Digitally Delivered Exercise and Education Treatment for Low Back Pain: 3 Months Follow-up
Acronym: Back3months
Status: Completed | Type: Observational
Sponsor: Joint Academy (Industry)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: Back study 3 months
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-05

CONDITIONS: Pain; Physical Function
Keywords: Low back pain; Pain; Exercise; Physiotherapy; Telehealth; Digital treatment
MeSH Terms: conditions — Pain; Low Back Pain; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Digitally delivered exercise and education treatment Joint Academy — The Joint Academy® (www.jointacademy.com) program for people with LBP consists of video instructed and progressively adaptable daily exercises, patient education through text lessons and a continuous asynchronous chat function with a personal reg. physiotherapist who supervises the patient during the full participation period. The program also contains three telephone consultations with a physiotherapist that were compulsory, one at the start, one after six weeks and one after three month.

SUMMARY:
Exercise and education is recommended as the first-line treatment by evidence-based, international guidelines for low back pain (LBP). Despite consensus regarding treatment, there is a gap between guidelines and what is offered to patients and less than half of the patients with nonspecific low back pain receive proper first-line care.

The aim of this study was to examine the short-term effect in pain and function in people with nonspecific LBP, participating in the digitally delivered treatment program Joint Academy.

DETAILED DESCRIPTION:
Low back pain (LBP) is the 4th leading cause of Disability Adjusted Life Years (DALYs) among adults aged 25-49.. According to evidence-based clinical guidelines, exercise and education constitute the first-line intervention. In an attempt to support the implementation of the guidelines, the BetterBack Modell of Care (MoC), a face-to-face concept including exercise and education, was developed and tested in primary care clinics in Sweden since 2017.

The BetterBack (MoC) is a package of education and training that includes structured assessment by a physiotherapist, information on cause and prognosis for LBP and individualised exercise. BetterBack has so far shown that physiotherapists experience increased self-efficacy for assessing and treating patients with LBP and that patients experience improved knowledge for self-care. Despite clinical guidelines for LBP, there is a gap between guidelines and what is offered to patients with LBP, and valuable health resources are still used for examinations and treatments that are proven ineffective or even harmful.

Traditional face-to-face interventions present barriers, such as limited access and lack of flexibility, which may limit the patients' adherence with the interventions. Digital delivery of the management program may be one way of overcoming such barriers. Telehealth, defined as the 'delivery of healthcare at a distance using information and communication technology' (ICT) could be a solution to many access barriers and has been rapidly adopted by many healthcare professions and accelerating even more throughout the COVID-19 pandemic.

Literature investigating the use of telehealth for the management of musculoskeletal pain is growing. Systematic reviews have demonstrated that telehealth can provide improvements in pain, physical function and disability that are similar to that of usual face-to-face care for individuals with musculoskeletal conditions such as osteoarthritis and non-specific low back pain. The use of telehealth also seems to increase exercise adherence for a variety of musculoskeletal conditions. However, there is a vast heterogeneity between studies included in these systematic reviews with respect to the intervention (type of exercise and education) and the ICT strategy provided, highlighting the need for further evidence-based digital programs to strengthen these findings.

Joint Academy® (JA), a digitally delivered treatment program with exercise and education was developed to increase access to and facilitate implementation of guideline derived and evidence-based treatment for musculoskeletal pain. The first JA program was introduced in 2016 for persons with hip- and knee OA and showed reduced pain and improved function. A recent randomized controlled trial on patients with knee OA showed that the digital program was superior to usual care. During 2021, a similar programme for persons with LBP, inspired by the Swedish face-to-face Better Back MoC was introduced.

The purpose of this study was to evaluate 3-months changes in pain and function during participation in the digitally delivered Joint Academy® (JA) exercise and education treatment program for patients with low back pain. A second aim was to examine the association of sociodemographis, health-related and treatment-related factors with outcome.

ELIGIBILITY:
Absolute exclusion criteria

* < age 18 years

  * Pregnancy
* Concerns of low back pain due to "red flags" (e. g cancer, fracture, infection, cauda equina syndrome)

Relative (to be further examined before inclusion)

* Radiculopati
* Previous or current cancer or unvoluntary weight loss
* Opioid demanding pain or pain in rest (cancer?, fracture?, infection?)
* Inflammatory back pain (atypical pain)
* Older patients (>75 years) with multiple disease
* Structural deformities (atypical pain)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants that have taken part of the digitally delivered treatment program for low back pain are reqruited from the Joint Academy database.
  Persons joined the program through recommendation by their local physiotherapist or via online advertisements and campaigns placed on search engines and social networks, or through their insurance company.
  A majority of included participants had a clinical diagnosis of non-specific LBP (diagnose code ICD-10 M54.5) from a PT or physician. Individuals without a prior diagnosis had a clinical diagnosis confirmed by a PT via telephone or videocall, or if deemed necessary be recommended to seek face-to-face care before inclusion in the programme.
Sampling Method: Non-Probability Sample
Enrollment: 2593 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale (NRS) | Weekly change from baseline to three months
  Pain was assessed weekly using the Numerical Rating Scale (NRS), with the instruction "Mark on this scale how much pain you had the last week in your hip/knee", followed by a 0-10 scale where 0 indicates No pain and 10 indicates Maximum pain.

SECONDARY OUTCOMES:
Oswersty Disability Index (ODI) | baseline and 3 months
  The ODI is divided into ten sections to assess the level of pain and interference with several activities including; sleep, self-care, sex life, social life and travelling. Each question has six possible responses which are scored from 0 to 5 (good to bad). The score for each section is added and divided by the total possible score (50 if all sections are completed), and the resulting score is multiplied by one hundred to yield a percentage score with 0% equivalent to no disability and 100% equivalent to a great deal of disability.
PASS | baseline and 3 months
  Patient Acceptable Symtom State, descriptive, not link to other patient-reported outcome measures. PASS was assessed at follow-up with the question: "Considering your lower back function, do you feel that your current state is satisfactory? (yes/no). The PASS is a treatment-response criterion developed to determine the clinical relevance of a treatment effect. Answering no is referred to as PASS(-), yes is referred to as PASS (+), and changing from no at baseline to yes at 3 months as PASS(-to+).
Radicular pain | baseline and 3 months
  Radicular pain assessed with Numerical Rating Scale (NRS), with the instruction "Mark on this scale how much pain you had the last week in your hip/knee", followed by a 0-10 scale where 0 indicates No pain and 10 indicates Maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Leif E Dahlberg, Senior professor, Study Director — Arthro Therapeutics /Joint Academy
Locations (1):
- Arthro Therapeutics, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be made available on request: either pseudonymized (coded) or aggregated original data, or of analyses performed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available when the paper has been submitted and accepted for publication and up to two years after that.
Access Criteria: Researchers can ask for access through contacting medical director and responsible researcher at Joint Academy.

REFERENCES:
- [Derived] Horder H, Nero H, Misini Ignjatovic M, Kiadaliri A, Lohmander LS, Dahlberg LE, Abbott A. Digitally Delivered Exercise and Education Treatment Program for Low Back Pain: Longitudinal Observational Cohort Study. JMIR Rehabil Assist Technol. 2022 Jun 21;9(2):e38084. doi: 10.2196/38084. PMID 35727622